CLINICAL TRIAL: NCT02708719
Title: Development of a Minimal Important Difference for the 1-minute Sit-to-stand Test
Brief Title: Development of a MID for the 1-minute Sit-to-stand Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MID 1-minute STST
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: COPD
Keywords: COPD; MID; 1-minute sit-to-stand-test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary rehabilitation (Other): multimodal pulmonary Rehabilitation program (3 weeks Duration)
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — Inpatient pulmonary rehabilitation has a duration of 3 weeks. This multimodal program consists of exercise training, breathing therapy, medical council, education and psychological support.

SUMMARY:
The purpose of this study is to determine the minimal important difference (MID) for the 1-minute-sit-to-stand-test (STST) with an anchor-based method.

DETAILED DESCRIPTION:
In this study we develop the minimal important difference for the 1-minute sit-to-stand-test (STST) with an anchor-based method.

First step of this study is to find out the differences in the number of repetitions during 1-minute STST, 6-minute walk distance and health-related quality of life from pre to post inpatient pulmonary Rehabilitation program (3 weeks Duration) in the Schoen-Klinik Berchtesgadener Land.

In Addition, Balance tests on the Leonardo-Mechanograph will be performed and the Hospital Anxiety and Depression Scale (HADS) and Chronic Respiratory Questionnaire (CRQ) will be assessed.

For the second step we will use an anchor-based approach to estimate the MID of the STST. 6MWD and CRQ are used as anchors for which the MID has been established before.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (GOLD-Stage II to IV)
* Ability to stand-up and walk
* written informed consent

Exclusion Criteria:

* orthopaedic or other comorbidities that prevent patients from performing the STST, 6MWT or exercise Training
* acute exacerbation
* heart failure, acute coronary syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
MID of the 1-minute-STST | 21 days
  Change of maximum 1-minute sit-to-stand repititions

SECONDARY OUTCOMES:
6-minute-walk distance | 21 days
  Maximal walk distance reached in 6 minutes
CRQ Score | 21 days
  CRQ is a health-related Quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Schoen Klinik BGL
Locations (1):
- Berchtesgardener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No